CLINICAL TRIAL: NCT02552862
Title: Study of the Effect of Adjunctive Vivomixx® in Addition to Antibiotics on Systemic and Cerebral Inflammatory Response in Patients With Cirrhosis and Spontaneous Bacterial Peritonitis (SBP)
Brief Title: Study of the Effect of Adjunctive Vivomixx® in Patients With Cirrhosis and Spontaneous Bacterial Peritonitis (SBP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No candidates during recruiting time. There were no candidates meeting the inclusion criteria
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-VSL-2014-49
Record Dates: First submitted 2015-08-26; First posted 2015-09-17 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vivomixx® (Active Comparator): Vivomixx® is a probiotic mixture of 8 proprietary strains. Thirty consecutive patients with cirrhosis and SBP will be randomized to receive Vivomixx® , sachets containing 450 x 109 bacteria, 2 every 12 hours during all the hospitalization until a maximum of 30 days (n=15), or placebo (n=15).
  All patients will receive endovenous antibiotics and also intravenous albumin 1.5 g/kg weight the first day and 1 g/kg weight the third day of treatment. The management of patients will follow current guidelines.
  Interventions: Drug: Vivomixx®
- Placebo (Placebo Comparator): Placebo will be formulated as identical in appearance and administered according to the same schedule as the active agent. Placebo contains maltose and silicon dioxide as inactive agent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vivomixx® — Vivomixx® is a probiotic mixture of 8 proprietary strains, namely Streptococcus thermophilus DSM 24731, bifidobacteria (B. breve DSM 24732, B. longum DSM 24736, B. infantis DSM 24737) and lactobacilli (L. paracasei DSM 24733, L. acidophilus DSM 24735, L. delbrueckii subsp bulgaricus DSM 24734, L. plantarum DSM 24730). The active agent will be supplied as a 4.4g sachet at a dose of 450 billion live bacteria per sachet with maltose and silicon dioxide as excipients.
  Other Names: Vivomixx ®
  Arms: Vivomixx®
Drug: Placebo — Placebo will be formulated as identical in appearance and administered according to the same schedule as the active agent. Placebo contains maltose and silicon dioxide as inactive agent.
  Arms: Placebo

SUMMARY:
Study Design: Double-blind placebo-controlled clinical trial

Study Duration:2 years

Study Center: Hospital de la Santa Creu i Sant Pau, Barcelona (single center)

Objectives: To assess the effect of adjunctive Vivomixx® on bacterial translocation in patients with cirrhosis and SBP

Number of Subjects: 30

Main Inclusion Criteria: Patients with cirrhosis hospitalized with an episode of SBP at Hospital de la Santa Creu i Sant Pau

Study Product, Dose, Route, Regimen: Vivomixx ® sachets containing 450 x 109 bacteria, 2 every 12 hours during hospitalization (n=15), or placebo (n=15)

Duration of administration: During hospitalization due to SBP episode

Hypothesis: The adjunctive treatment with Vivomixx® in patients with cirrhosis and SBP could decrease bacterial translocation and systemic and cerebral proinflammatory state. This would result in a faster SBP resolution, a decrease in the incidence of complications and an improvement in cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis hospitalized with an episode of SBP at Hospital de la Santa Creu i Sant Pau.

Cirrhosis will be diagnosed by clinical, analytical and ultrasonographic findings or by liver biopsy. SBP will be diagnosed by an ascitic fluid neutrophil count > 250/mm3 with or without positive culture .

Exclusion Criteria:

* Advanced hepatocellular carcinoma (beyond Milan's criteria) or any other malignancy.
* Advanced liver insufficiency [MELD (model for end-stage liver disease) >25].
* Active alcohol intake (in the previous 3 months).
* Neurological disease.
* Marked symptomatic comorbidities (cardiac, pulmonary, renal, untreated active depression, HIV infection).
* Previous antibiotic treatment, including norfloxacin and rifaximin.
* Septic shock, ileus, need for tracheal intubation or intensive care unit.
* Immunomodulatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in bacterial translocation (composite measure) | At baseline, daily until infection resolution (an expected average of 7 days) and at three months after discharge
  Bacterial translocation will be evaluated by change from baseline in bacterial DNA in blood and ascitic fluid, lipopolysaccharide binding protein (LBP), intestinal fatty acid-binding protein (I-FABP) and intestinal bile acid binding protein (I-BABP) in blood, and polyethylene glycols (PEG) and claudin 3 in urine .

SECONDARY OUTCOMES:
Changes in systemic inflammatory response and systemic oxidative damage (composite measure) | At baseline, daily until infection resolution (an expected average of 7 days) and at three months after discharge
  Systemic Inflammation and immune response will be evaluated by change from baseline in serum C reactive protein (CRP), interleukin (IL)-1β, IL-6, tumor necrosis factor (TNF)-α, IL-10, IL-12, IL-18, IL-22, sTNFR-1, sTNFR-2, sCD163, matrix metalloproteinase (MMP) -9, interferon (IFN)-γ, vascular endothelial growth factor (VEGF), claudin-5, nitrites and nitrates in serum and ascitic fluid.
  Systemic oxidative damage will be evaluated by change from baseline in determination of malondialdehyde (MDA) in blood.
Changes in cognitive function (composite measure) | At baseline at infection resolution (an expected average of 7 days)
  Cognitive function will be evaluated by change from baseline in Trail-Making Test A (TMT-A), Trail-Making Test B (TMT-B), and Digit Symbol Test (DST).
Changes in brain inflammation (composite measure) | At baseline (during the first 12-24 hours after inclusion in the study) and after 3 days of treatment.
  Brain inflammation will be evaluated by change from baseline in MRI and different biomarkers of neuroinflammation.
  A designed MR protocol will be produced, including imaging using different sequences, and more biochemical (MR spectroscopy) and functional (DTI) studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain